CLINICAL TRIAL: NCT03497442
Title: Treatment of Asian Flushing Syndrome With Topical Alpha Agonists
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 17-23964
Record Dates: First submitted 2018-04-05; First posted 2018-04-13 (Actual); Last update posted 2020-05-04 (Actual); Status verified 2020-04

CONDITIONS: Flushing; Alcohol-Related Disorders; Aldehyde Dehydrogenase Deficiency
MeSH Terms: conditions — Flushing; Alcohol-Related Disorders | interventions — Brimonidine Tartrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a split face study. All participants will follow an identical protocol with active medication applied to half of their face and placebo applied to the other half. Treatment and placebo side will be randomized.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Treatment Arm (Experimental): This is a randomized vehicle controlled, double blinded, interventional study. Patients of East Asian descent with a history of Asian Flushing Syndrome will be asked to apply a thin layer of brimonidine 0.33% gel to one half of their face thirty minutes before consuming alcohol (1.5 oz vodka for women, 3.0 oz vodka for men). The Photos will be taken 30 minutes, one hour, and 1.5 hours after consumption of alcohol. Erythema will be assessed at each time point by both the patient and study investigator using a 5- point erythema assesment score. Patient blood alcohol content (BAC) will be measured noninvasively at each time point.
  Interventions: Drug: Brimonidine Tartrate
- Placebo Arm (Placebo Comparator): This is a randomized vehicle controlled, double blinded, interventional study. Patients of East Asian descent with a history of Asian Flushing Syndrome will be asked to apply a thin layer of vehicle gel to one half of their face thirty minutes before consuming alcohol (1.5 oz vodka for women, 3.0 oz vodka for men). The Photos will be taken 30 minutes, one hour, and 1.5 hours after consumption of alcohol. Erythema will be assessed at each time point by both the patient and study investigator using a 5- point erythema assesment score. Patient blood alcohol content (BAC) will be measured noninvasively at each time point.
  Interventions: Drug: Placebo Vehicle Gel

INTERVENTIONS:
Drug: Brimonidine Tartrate — Topical brimonidine tartrate will be applied to one half of each participant's face. A randomization process will be used to determine which side of the face each participant will apply treatment to. The untreated side of the face will receive a placebo vehicle. Patient and clinician will be blinded to treatment side.
  Other Names: Mirvaso
  Arms: Treatment Arm
Drug: Placebo Vehicle Gel — Vehicle Gel
  Arms: Placebo Arm

SUMMARY:
Asian Flushing Syndrome (AFS) is a genetic disease affecting approximately 70% of patients of East Asian descent characterized by severe flushing with minimal ethanol consumption. This reaction is cosmetically unattractive and socially limiting. Many Asian patients avoid drinking alcohol on dates, at weddings, and during business events because of this reaction and the perception of being drunk or alcoholic.

Ethanol is normally metabolized to acetic acid by two enzymes. The first enzyme, alcohol dehydrogenase (ADH) converts ethanol to acetaldehyde. The second enzyme, aldehyde dehydrogenase 2 (ALDH2) converts the toxic acetaldehyde to harmless acetic acid. When ADH function is increased or ALDH2 function is decreased, the toxic intermediate acetaldehyde accumulates resulting in cutaneous flushing. Over 70% of East Asians have genetic polymorphisms in either ADH or ALDH2 leading to intense flushing with ethanol consumption.

There are no effective topical treatments for the Asian Flushing Syndrome. Oral antihistamines have been used with some success in treating symptoms of Asian Flushing Syndrome; however these can have sedating effects and may be dangerous in combination with alcohol.

Brimonidine is a selective α2-adrenoceptor agonist that acts through vasoconstriction and is commercially available in a topical gel. This topical treatment is FDA approved for the indication of facial flushing and has a long history of safety in human subjects.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 21 years of age or older
* Self-reported East Asian descent defined as being at least partially ethnically Han Chinese, Japanese, or Korean.
* No persistent facial erythema at baseline as reported by the patient and observed by investigators at first visit
* Moderate to severe facial erythema (grade of 2 or more on the Clinician Erythema Assessment scale) induced by one standard drink of alcohol as defined by the National Institute on Alcohol Abuse and Alcoholism (12 ounces of beer, 5% alcohol; 5 ounces of wine, 12% alcohol; or 1.5 ounces of distilled spirits, 40% alcohol). Patients must provide a photo of themselves in sufficient lighting after having one standard drink to be confirmed by the investigators at the screening visit.
* Written informed consent for any and all study procedures
* Written authorization for use and release of health and research study information
* Written authorization for use of photos in publications and presentations
* Ability to follow study instructions and complete study assessment tools without assistance.
* Ability to communicate with the study team without the need for translators.
* Female patients of childbearing potential must have a negative urine pregnancy test result at the screening visit.

Exclusion Criteria:

* Age < 21
* Known hypersensitivity or allergies to any component of the study treatment
* Pregnancy or active breastfeeding
* History of rosacea
* Exam findings consistent with rosacea
* Current use of medications for rosacea
* Current use of oral H1 or H2 antagonists, or use in the last 2 weeks
* Active acne vulgaris
* Current use of topical medications for acne vulgaris
* Any uncontrolled systemic disease or abnormal vital signs at study visit
* Current use of medications known to cause cutaneous flushing such as rifampin, nicotinic acid, calcium channel blockers (or other antihypertensives), nitroglycerin, prostaglandins, bromocriptine, tamoxifen, thyroid hormone replacement, cyproterone acetate (or other medications to induce fertility), sildenafil citrate, and monoamine oxidase inhibitors
* Current use of medications known to be contraindicated with alcohol use such as disulfiram, rifampin, isoniazid, isotretinoin, anxiolytics, non-steroidal anti-inflammatory medications, acetaminophen, warfarin, antidepressants, St. John's Wort, cyclobenzaprine and other muscle relaxants, metronidazole, trimethoprim-sulfamethoxazole.
* History of any of the following conditions: Raynaud's syndrome, orthostatic hypotension, cerebral or coronary insufficiency, congenital or acquired heart disease, thromboangiitis obliterans, alcohol or substance abuse, liver fibrosis or cirrhosis, hepatitis, renal insufficiency, severe gastrointestinal bleeding, seizures, or psychiatric disease.
* Protected or vulnerable patient groups such as inmates, children and minors, pregnant women, and individuals with cognitive impairment or those who are legally blind, illiterate, or cannot talk or write.
* Use of any products containing oxymetazoline or brimonidine within 2 weeks of initial study visit.
* Use of topical glucocorticosteroids applied to the face within 2 weeks of initial study visit
* Any prior treatment with lasers, intense pulsed light, photodynamic therapy, or other energy based therapy to the face.
* Facial hair, tattoos, facial characteristics, or cutaneous disease (such as actinic damage, melasma, postinflammatory hyper- or hypopigmentation, excessive telangiectasias, nevi, or other pigmentation) which may interfere with assessments of erythema in the opinion of the investigators.
* Current enrollment in an investigational drug or device study or participation in such within 30 days of entry into this study.
* Any condition or situation that, in the investigator's opinion, may put the patient at significant risk, or may significantly interfere with the patient's participation in the study.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-07-12 (Actual); Primary Completion 2019-03-25 (Actual); Study Completion 2019-03-25 (Actual)

PRIMARY OUTCOMES:
Clinician Erythema Score | Evaluated 30 minutes after alcohol consumption
  Clinician Erythema Assessment (CEA) Scale Grade 0: Clear skin with no signs of erythema Grade 1: Almost clear of erythema, slight redness Grade 2: Mild erythema, definite redness Grade 3: Moderate erythema, marked redness Grade 4: Severe erythema, fiery redness.
Patient Erythema Self Assessment | Evaluated 30 minutes after alcohol consumption
  Subject self-assessment 0: No signs of unwanted redness
  1. Almost clear of unwanted redness
  2. Mild redness
  3. Moderate redness
  4. Severe redness

SECONDARY OUTCOMES:
Delayed Clinician Erythema Score | Evaluated 60 and 90 minutes after alcohol consumption
  Clinician Erythema Assessment (CEA) Scale
Delayed Patient Erythema Self Assessment | Evaluated 60 and 90 minutes after alcohol consumption
  Subject self-assessment

CONTACTS AND LOCATIONS:
Overall Officials: Wesley Yu, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- UC, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brooks PJ, Enoch MA, Goldman D, Li TK, Yokoyama A. The alcohol flushing response: an unrecognized risk factor for esophageal cancer from alcohol consumption. PLoS Med. 2009 Mar 24;6(3):e50. doi: 10.1371/journal.pmed.1000050. PMID 19320537
- [Background] Eng MY, Luczak SE, Wall TL. ALDH2, ADH1B, and ADH1C genotypes in Asians: a literature review. Alcohol Res Health. 2007;30(1):22-7. PMID 17718397
- [Background] Miller NS, Goodwin DW, Jones FC, Gabrielli WF, Pardo MP, Anand MM, Hall TB. Antihistamine blockade of alcohol-induced flushing in orientals. J Stud Alcohol. 1988 Jan;49(1):16-20. doi: 10.15288/jsa.1988.49.16. PMID 3347071
- [Background] Altura BM, Carella A, Altura BT. Acetaldehyde on vascular smooth muscle: possible role in vasodilator action of ethanol. Eur J Pharmacol. 1978 Nov 1;52(1):73-83. doi: 10.1016/0014-2999(78)90023-7. PMID 720389
- [Derived] Yu WY, Lu B, Tan D, Aroyan C, Shinkai K, Leslie KS, Fox LP, Yu S, Neuhaus IM, Grekin RC, Arron ST. Effect of Topical Brimonidine on Alcohol-Induced Flushing in Asian Individuals: A Randomized Clinical Trial. JAMA Dermatol. 2020 Feb 1;156(2):182-185. doi: 10.1001/jamadermatol.2019.3508. PMID 31799996